CLINICAL TRIAL: NCT06434129
Title: Role of Diffusion Tensor-magnetic Resonance Imaging in Investigating Sensorineural Hearing Loss
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohammad Aly, Assistant lecturer, Assiut University
Other Study IDs: 1a
Record Dates: First submitted 2024-05-21; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Sensorineural Hearing Loss
Keywords: DTI; Sensorineural hearing loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: cases with SNHL
  Interventions: Diagnostic Test: DTI
- Controls: Normal people
  Interventions: Diagnostic Test: DTI

INTERVENTIONS:
Diagnostic Test: DTI — Diffusion MRI imaging

SUMMARY:
DTI and auditory tractography can be incorporated into the diagnostic toolkit for patients who are scheduled to undergo cochlear implantation and whose standard assessments have been unable to determine the functional integrity of the auditory pathway. These techniques aid in decision-making processes regarding potential outcomes, determining the optimal side for implantation, providing counseling regarding the possibility of limited benefits from surgery, and considering alternative forms of rehabilitation. The investigators including patients with varying degrees of hearing loss, as well as patients with normal radiological findings who are scheduled for cochlear implantation. The ultimate goal is to create a comprehensive map across the entire hearing spectrum and validate the findings of this study..

DETAILED DESCRIPTION:
Hearing is a complex process in which many parts of the ear contribute to transmit signals to the brain. The auditory system consists of both peripheral structures (external, middle, and inner ear)as well as central regions (cochlear nuclei in the medulla oblongata, superior olivary nuclei and lateral lemniscus in the pons, inferior colliculus in the midbrain, medial geniculate nuclei in the thalamus, and auditory cortex in the superior temporal Heschl gyrus). Most of auditory fibres undergo a contralateral decussation to the opposite superior olive in the region known as the trapezoid body.

The broad term "sensorineural hearing loss" (SNHL) It accounts for a substantial proportion of hearing impairment cases globally, affecting individuals of various age groups. It has been used by clinicians to refer to either malfunctioning inner ear or a retrocochlear problem affecting the canalicular vestibule-chochlear (VIII) cranial nerve and cerebellopontine angle or that involves the higher (central) auditory nuclei and neural tracts. Identifying the etiology of hearing loss is valuable to establish a treatment strategy that can help to prevent or slow down complete loss of auditory function.

The central auditory structures are involved in various processes that may occur in isolation from those involving peripheral receptors .SNHL can be a consequence of different conditions, including viral infection, tumor, ischemia, multiple sclerosis, or congenital malformations.

Despite continuous efforts to delineate the pathophysiological attributes of SNHL, the aetiology remains mostly unclear with nearly 90% of cases being idiopathic. Therefore, finding a method to accurately predict microstructural changes of the auditory circuit is extremely important.

Conventional imaging modalities, including computed tomography (CT) and magnetic resonance imaging (MRI), have offered invaluable insights into the macroscopic changes associated with SNHL, such as cochlear morphology and structural abnormalities. However, these techniques lack the sensitivity to discern subtle alterations occurring at the microstructural level, impeding a comprehensive understanding of the underlying pathophysiological processes.

DTI-MRI's ability to capture subtle changes in tissue microstructure makes it an ideal candidate for probing the intricate auditory pathways affected by SNHL. By quantifying the diffusion of water molecules along axonal pathways, DTI-MRI can uncover alterations in the integrity of auditory neural connections, which are often missed by conventional imaging methods. Furthermore, DTI-derived metrics, such as fractional anisotropy (FA), axial diffusivity (AD), radial diffusivity (RD), and mean diffusivity (MD), offer quantitative measures to characterize the white matter integrity and myelination in auditory pathways.

ELIGIBILITY:
Inclusion Criteria:

* Patients with audiometrically proven SNHL

Exclusion Criteria:

* Neurologically or psychiatric conditions affecting patient stability during MRI examination.
* Cochlear implants.
* Contraindications for MRI.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Assiut university hospital patients
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of role of DTI in SNHL | one year
  Assess the integrity of auditory pathway via measuring DTI metrics ( Fractional anisotropy and mean diffusivity)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine of Assuit, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided